CLINICAL TRIAL: NCT00242112
Title: Defining the Extent and Grade of Prostate Cancer Using Dynamic Contrast Enhanced Diffusion Weighted and BOLD MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-0387-CE
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- MRI - pathology (Other)
  Interventions: Procedure: MRI Prostate

INTERVENTIONS:
Procedure: MRI Prostate

SUMMARY:
The purpose of this study is to determine the ability of functional MRI techniques to detect, measure and locate intra-prostatic cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine the ability of functional MRI techniques [High Resolution Dynamic Contrast Enhanced MRI (HR-DCE-MRI), diffusion weighted MRI (DWI) and BOLD MRI] to detect, measure and locate intra-prostatic cancer. 70 patients undergoing MRI for staging of prostate cancer prior to radical prostatectomy will be studied. Results of MRI obtained prior to surgery will be correlated with pathologic specimens to determine MRI accuracy.

ELIGIBILITY:
Patients will be recruited from the University Health Network (UHN). Eligible patients will be undergoing radical prostatectomy for prostate cancer at UHN. Patients with a contraindication to MRI or MRI contrast agents, claustrophobia, renal failure, allergy to MRI contrast agents, or prior hormonal therapy or radiation therapy for prostate cancer, a biopsy within 3 weeks of the surgical date or active prostatitis will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Extent and Grade of Prostate Cancer Using MRI | Imaging followed by pathology analysis
  Before undergoing surgery, all patients were examined with MR imaging

CONTACTS AND LOCATIONS:
Overall Officials: Masoom Haider, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada